CLINICAL TRIAL: NCT06558383
Title: Augmented Posterior Oblique Sling Activation on Lumbopelvic Recruitment Pattern and Functional Outcomes in Lumbosacral Radiculopathy Patients
Brief Title: Augmented Posterior Oblique Sling Activation on Lumbopelvic Recruitment Pattern in Lumbosacral Radiculopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Refaat Kamal, assistant lecturer of physical therapy for neurology and neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005233
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Lumbosacral Radiculopathy
Keywords: posterior oblique sling; recruitment pattern; lumbar radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. True experimental research design study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group - (Active Comparator): Control group (A):
  Twenty patients will receive selected physical therapy program for 18 sessions, three sessions per week for six weeks in form hot packs, soft tissue techniques, mobilization and manipulation of lumbar spine, and neurodynamics.
  Interventions: Other: selected physical therapy program
- study group (Active Comparator): Study group (B):
  Twenty patients will receive augmented activation of posterior oblique sling in addition to selected physical therapy program, 18 sessions, three sessions per week for six week
  Interventions: Other: augmented posterior oblique sling activation; Other: selected physical therapy program

INTERVENTIONS:
Other: augmented posterior oblique sling activation — activation of posterior oblique sling for 18 sessions, three sessions per week for six weeks
  Arms: study group
Other: selected physical therapy program — selected physical therapy program for 18 sessions, three sessions per week for six weeks in form hot packs, soft tissue techniques, mobilization and manipulation of lumbar spine, and neurodynamics and stabilization exercises

SUMMARY:
The current study aims to determine the impact of augmented posterior oblique sling activation on lumbopelvic recruitment pattern and functional outcomes in patients with unilateral lumbosacral radiculopathy.

DETAILED DESCRIPTION:
Low back pain is now the leading cause of disability worldwide. Back pain and its related disability have a huge impact on individuals, communities, and healthcare systems. It reduces an individual's ability to participate in work which in turn negatively affects their quality of life. Also, it has major economic consequences through increasing the cost of health care and work absenteeism. Among the many differentials of low back pain, the most common cause is lumbosacral radiculopathy. Patients with low back pain showed uncontrolled lumbopelvic mobility while performing hip extension movement in functional activities. In patients with back pain, there is over-activation of the hamstrings and erector spinae and delayed or absent contraction of the gluteus maximus. Clinically, this pattern is observed as an anterior pelvic tilt with increased extension in the lumbar spine as the patient lifts the leg into extension. So, repetition of this abnormal pattern in patients with lumbosacral radiculopathy may result in mechanical and compressive stresses in the lumbar spine and magnify the patient's symptoms. Despite the role of POSM in improving spinal mobility and stability. And stabilizing the lumbopelvic joint, there are no previous studies investigating the impact of activation posterior oblique activation on this abnormal lumbopelvic recruitment and functional outcomes in patients with lumbosacral radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 25 to 40
* L4/5 and L5/S1 disc herniation.
* Duration of pain will be more than three months.
* Normal body mass index (18.5 - 24.99Kg/m2)

Exclusion Criteria:

* 1. Red flags: spinal tumors, cauda equina syndrome, spinal fractures, osteoporosis, infection.

  2. Bilateral symptoms. 3. Spondylolisthesis, spondylitis, and spinal canal stenosis. 4. Previous lumbopelvic or hip surgery or injection 5. Any hip structural abnormality such as malformations, impingements and degeneration.

  6. Postural deviations such as scoliosis, kyphosis, lateral shift. 7. True leg length discrepancy. 8. Pregnancy and Gynecological problems.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
surface EMG unit | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  The electromyographic pattern of activation of lumbopelvic musculature (sequence and level of activity) will be measured during prone hip extension testing using surface EMG unit.
Pressure biofeedback unit | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  it will be used to assess pelvic motion. the pressure sensor of the pressure biofeedback unit will be placed anteriorly between the patients' ilium and the testing table. The amount of pressure applied by the patient on the sensor at rest will be recorded then, the amount of pressure applied by patients at prone hip extension at 10 degrees will be recorded.

SECONDARY OUTCOMES:
pressure algometry | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  The pressure algometry will used to measure pressure pain threshold in low back area and in sciatic valleix.
Arabic version of Oswestry Low Back Pain Disability Questionnaire | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  back pain-related disability will be assessed using using the Arabic version of Oswestry Low Back Pain Disability Questionnaire.It is a 10-item self-reported questionnaire. The patient will be asked to answer every question and mark only the box that most closely describes his problem. Each question will be assessed on a six-point scale ranging from 0 (no disability) to 5 (major disability). The score is determined by adding each item score together. The overall score is out of 50 . Higher scores represent greater disability.
back pain intensity using the Visual analogue scale | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  The subject will be asked to make a handwritten mark on a 100 mm line (10cm). This line represents a continuum between no pain or discomfort (zero), and the worst pain (10) the patient could feel. Measurements from the starting point of the scale to the patients' marks will be recorded and interpreted as their pain intensity. Higher scores represent greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda M Zakaria, professor, Study Chair — Cairo University; Ebtesam M Fahmy, professor, Study Chair — Cairo University; Nagwa M Ibrahim, Study Chair — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No